CLINICAL TRIAL: NCT05723809
Title: Treatment of Lateral Epicondylitis With a Percussive Therapy Device: Outcomes of a Randomized Controlled Trial
Brief Title: Treatment of Lateral Epicondylitis With a Percussive Therapy Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Therabody, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Stone, Principal Investigator, Assistant Professor, Orthopedic Surgeon, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002285
Record Dates: First submitted 2023-01-30; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Percussive Therapy Device (Experimental): Participants will be going to physical therapy - 1 session per week for 6 weeks and will use a percussive therapy device daily for 3-7 minutes
  Interventions: Device: Percussive Therapy Device; Behavioral: Physical Therapy
- Control group (Active Comparator): Participants will be going to physical therapy - 1 session per week for 6 weeks
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Device: Percussive Therapy Device — Same as group description
  Other Names: Theragun
  Arms: Percussive Therapy Device
Behavioral: Physical Therapy — Same as group description

SUMMARY:
The purpose of this study is to assess the efficacy of using a percussive therapy device in addition to physical therapy to treat acute tennis elbow

DETAILED DESCRIPTION:
The device the investigators intend to use is Class I and in a class of devices that is exempt from the FDA requirement for premarket notification/approval (exempt from 510K or PMA), which would not be "subject to section 510(k), 515, or 520(m) of the Federal Food, Drug, and Cosmetic Act" (ref: FDAAA Checklist)

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older are included
* Patients with atraumatic lateral epicondylitis symptoms
* Symptoms persistent and present for at least 2 weeks
* Presence of 2 of the following on clinical examination: +tenderness to palpation common extensor tendons and/or lateral epicondyle origin, pain over the lateral elbow with passive flexion of the wrist in an extended position, +pain with resisted supination, +pain with resisted middle finger extension.

Exclusion Criteria:

* Any records flagged "break the glass" or "research opt out."
* Patients with elbow osteoarthritis,
* Patients with a history of traumatic injury to the elbow
* Patients with workers compensation
* Patients who received cortisol injection in the elbow
* MRI evidence of common extensor tear
* A history of surgery on the affected elbow,
* Cognitive or behavioral problems which would preclude informed consent.
* Patients with coagulopathies
* Patients who are pregnant
* Patients who had a cortisone injection within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to Improvement of Symptoms | 3 months

SECONDARY OUTCOMES:
PROMIS Upper Extremity | 3 months
  Patient-Reported Outcomes Measurement Information System
  Upper extremity - 0-100 indicating functionality of the upper extremity with higher scores representing more functionality
PROMIS Physical Functioning | 3 months
  Patient-Reported Outcomes Measurement Information System
  Physical function 0-100 indicating overall functionality with higher scores representing more functionality
PROMIS Pain Interference | 3 months
  Patient-Reported Outcomes Measurement Information System
  Pain interference 0-100 measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities with higher scores representing more interference
PROMIS Depression | 3 months
  Patient-Reported Outcomes Measurement Information System
  Depression - 0-100 assess self-reported negative mood (sadness, guilt), views of self (self- criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose) with higher scores indicating more depression
VAS pain score | 3 months
  Visual Analog Score for pain - subjective measure for acute and chronic pain. Scaled 0-10
SANE score | 3 months
  Single Assessment Numeric Evaluation - This is a single-question outcome measure that asks patients to rate their function, as it pertains to the area being treated, on a scale of 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Stone, M.D, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No